CLINICAL TRIAL: NCT02764515
Title: Comparison of the Efficacy and Safety of Kunxian Capsule and Methotrexate for the Treatment of Rheumatoid Arthritis
Brief Title: Kunxian for the Treatment of Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese SLE Treatment And Research Group (Other)
Collaborators: CHENLIJI Pharmaceutical Company,Guangzhou Pharmaceutical Group (Unknown); CHINESE RHEUMATISM DATA CENTER (Unknown)
Responsible Party: Principal Investigator, Xinping Tian, MD, Chinese SLE Treatment And Research Group
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Chenliji001
Record Dates: First submitted 2016-03-26; First posted 2016-05-06 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Kunxian Capsule; efficacy; rheumatoid arthritis; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — kunxian; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kunxian capsule group (Experimental): Intervention:
  Drug: Kunxian 2 capsules BID taken by mouth for 24 weeks. Kunxian capsule is composed of 4 ingredients: Tripterygium wilfordii Hook F 300mg, extracts from Gouqizi,Tusizi and yinyanghuo.
  Interventions: Drug: Kunxian Capsule
- Methotrexate group (Active Comparator): Intervention:
  Drug: Methotrexate tablet 10mg taken by mouth every week for 24 weeks.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Kunxian Capsule — Patients in the Kunxian Capsule group will take Kunxian Capsule 0.6gm orally twice daily for 24weeks
  Other Names: Tripterygium wilfordii Hook F.
  Arms: Kunxian capsule group
Drug: Methotrexate — the Methotrexate group will take Methotrexate 10mg orally every week for 24 weeks
  Other Names: jiaandieling
  Arms: Methotrexate group

SUMMARY:
This is a multicenter, randomized, double blind, double-dummy and controlled clinical trial aimed to compare the clinical efficacy and safety of Kunxian Capsule, a compound of Chinese traditional medicine, and the active comparator,Methotrexate for the treatment of rheumatoid arthritis. The primary end-point is that Kunxian Capsule is not inferior to Methotrexate both in efficacy and safety.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double blind, double-dummy and controlled clinical trial.The goal is to compare the clinical efficacy and safety of Kunxian Capsule, a compound of 4 ingredients of Chinese herb-derived medication, and the active comparator, Methotrexate for the treatment of mild to moderate active rheumatoid arthritis.This study is basically non-inferiority in design, so 428 subjects will be enrolled. All subjects need to fulfill the inclusion criteria and without exclusion criteria. Subjects are randomized into the Kunxian Capsule treatment group and Methotrexate treatment group.The dosage of Kunxian Capsule used in this study is 0.6g twice daily and the methotrexate dosage is 10mg per week. All subjects will take the medication for 24 weeks. Diclofenic is used as the salvage therapy in case patients experience joint pain. The primary end-point is the proportion of patients who could achieve disease remission or low disease activity treated with Kunxian Capsule and Methotrexate. All patients will be followed at week 2,4,12 and 24 after screening. Baseline information for disease activity measures such as DAS28 score,CDAI score, SDAI score, ACR20, ACR50, ACR70 improvement, HAQ score, patient's VAS score for pain, and lab tests such as CRP, ESR, RF, CCP, blood and urine routine tests, liver as well as renal function tests were collected and recorded. All these measures are performed at each follow-up visit except RF and CCP. In addition, any adverse events or withdrawal happened during each visit will be recorded for data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who understand the study protocol and sign the informed consent；
2. Fulfill the 1987 or 2010 ACR classification criteria for RA；
3. Male or female patients, age ranged from 40-70;
4. Male or female who do not plan to have more child,or per-menopausal or menopausal women；
5. Patients with mild or moderate disease activity, ie, whose DAS28 ranged from 3.2-5.1（ie, ESR>28mm/h，or patients who have 1-5 swollen joints as well as 1-5 tender joints）；
6. Without severe systemic disorders,such as severe pericardial effusion,pulmonary interstitial fibrosis,renal tubual acidosis,atrophic gastritis,autoimmune liver disease etc.
7. Not included in any drug trial 1 month before enrollment

Exclusion Criteria:

1. Pregnant woman or women who are preparing to pregnant or breast feeding；
2. Patients with active liver diseases or elevated liver enzymes eg, the ALT and/or AST is higher than 1.5 of the upper limit of normal range;
3. Patients with renal function abnormality,eg,serum creatinin higher than the upper limit of normal range；
4. White blood cell count less than 3.0×109/L，or with anemia(hemoglobin level lower than 80g/L），or platelet count less than 80×109/L，or with other hematological diseases;
5. Patients with chronic gastrointestinal diseases；
6. Patients with un-controlled hypertension,metabolic diseases such as diabetes;
7. History of malignant tumor or has malignant tumor at present;
8. With acute and/or chronic contagious diseases；
9. Severe arrhythmia on ECG test;
10. History of adverse reaction with Kunxian capsule,or Tripterygium wilfordii Hook F.,methotrexate or medications contain kunminshanhaitang ingredient；
11. History of psychiatric diseases or alcoholism or drug abuse；
12. Having been diagnosed to have systemic rheumatic diseases;
13. Ever taken immunosuppressive agents or biological agents or Tripterygium wilfordii Hook F or medications contain kunminshanhaitang ingredient in recent 3 months；
14. Had ever taken methotrexate or Kunxian capsule for more than 12 weeks but could not control the arthritis under remission；
15. With other conditions that are considered to be inconsistent with the inclusion criteria according to the investigators.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with ACR 20/50/70 | 24 weeks from baseline
  the percentage of patients who have ACR 20,50 and 70 treatment response after treated with Kunxian Capsule and Methotrexate for 24 weeks

SECONDARY OUTCOMES:
Proportion of patients whose DAS28 score less than 2.6 or 3.2 after treated with Kunxian Capsule and Methotrexate | 24 weeks from baseline
  Percentage of patients whose DAS28 could be lower than 3.2 or 2.6 after treated with Kunxian Capsule and Methotrexate for 24 weeks
Proportion of patients with adverse events in the Kunxian Capsule treatment group | 24 weeks from baseline
  The adverse events profile such as gastrointestinal tract adverse events, the percentage of patients with gonodal gland toxicities, liver function abnormalities, hematological abnormalities,skin rashes etc in patients treated with Kunxian Capsule will be analyzed and compared with the adverse events in patients treated with Methotrexate during the same time period.

CONTACTS AND LOCATIONS:
Overall Officials: XIAOFENG ZENG, MD, Principal Investigator — Peking Union Medical College Hospital; XINPING TIAN, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (16):
- China (16):
  - the Affiliated Hospital to Bangbu Medical University, Bengbu, Anhui
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - AnHui provincial hospital, Hefei, Anhui
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Third Affiliated Hospital to SUN YAT-SEN University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Harbin Medcial University, Haerbin, Heilongjiang
  - The first affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - Minda Hospital of Hubei Province, Enshi, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Xijing Hospital, Xian, Shanxi
  - the Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Guang'anmen Hospital,China Academy of Chinese Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Guang Hua hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No